CLINICAL TRIAL: NCT02201212
Title: A Phase II Trial of Everolimus for Cancer Patients With Inactivating Mutations in TSC1 or TSC2 or Activating MTOR Mutations
Brief Title: Everolimus for Cancer With TSC1 or TSC2 Mutation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, David Kwiatkowski, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-229; CRAD001MUS217T
Record Dates: First submitted 2014-07-23; First posted 2014-07-28 (Estimated); Results first posted 2020-09-16 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: TSC1; TSC2; Tuberous Sclerosis Complex; MTOR
Keywords: TSC1; TSC2; Tuberous Sclerosis Complex; MTOR
MeSH Terms: conditions — Tuberous Sclerosis | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Everolimus (Experimental): Everolimus
  * Fixed doses orally once a day per each 28 day cycle
  * Participants will stay on study as long as they do not progress for a maximum of 24 months.
  * Tumor assessments will be performed after every 2 cycles for as long as they are on study.
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus
  Other Names: Afinitor®; Zortress; Afinitor Disperz®; RAD001

SUMMARY:
In this research study, the investigators are evaluating the clinical benefit of everolimus in cancer patients with inactivating TSC1 or TSC2 mutations or activating MTOR mutations.

This research study is a Phase II clinical trial, which tests the safety and effectiveness of an investigational drug called everolimus to learn whether the drug works in treating a specific cancer. "Investigational" means that the drug is being studied. It also means that the FDA (the U.S. Food and Drug Administration) has not yet approved everolimus for your type of cancer.

Everolimus is a drug that may stop cancer cells from growing by blocking an important factor (mTOR) involved in the growth of cells. This drug has been used in treatment for other cancers and is approved by the Food and Drug Administration for treatment of several types of cancer, including renal cell carcinoma. Treatment with this drug has been associated with responses in some patients whose cancers had mutations in TSC1 or TSC2. The investigators think that patients whose tumors have mutations in TSC1 or TSC2 may have a good chance of responding to treatment with drugs like everolimus.

DETAILED DESCRIPTION:
Patients who fulfill eligibility criteria will be entered into the trial.The participant will be given a study drug-dosing calendar for each treatment cycle. Each treatment cycle lasts 28 days (4 weeks), during which time the participant will be taking the study drug orally (by mouth) once daily. The diary will also include special instructions for taking the study drug. In addition to the administration of the study drugs the participant will be asked to return to the clinic at various time points so that additional exams can be performed. These study visits may last as long as 2 hours.

ELIGIBILITY:
Inclusion Criteria: Participants must meet the following criteria on screening examination to be eligible to participate in the study:

* Participants must have histologically confirmed advanced malignancy that is either metastatic and/or unresectable and/or recurrent, with confirmed inactivating mutations in TSC1 or TSC2, or activating mutations in MTOR, identified in any CLIA-certified laboratory. All genetic findings must be reviewed by the study PI, Dr. David Kwiatkowski, prior to study entry.
* Biopsy of a primary or metastatic lesion must have been performed within the past two years. Sufficient pathologic material must be available to enable whole exome sequencing at the time of study entry.
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 20 mm with conventional techniques or as ≥10 mm with spiral CT scan. See section 10 for the evaluation of measureable disease.
* Participants may have received any number of prior therapies, from 0 to > 10, but prior treatment with PI3-kinase or mTOR inhibitors is not permitted.
* Age ≥ 18 years.
* ECOG performance status <2 (see Appendix A).
* Participants must have normal organ and marrow function as defined below:

  * Leukocytes ≥3,000/mcL
  * Absolute neutrophil count ≥1,500/mcL
  * Platelets ≥100,000/mcL
  * Hemoglobin ≥9.0 gr/dL
  * Total bilirubin ≤1.5 ULN
  * AST (SGOT)/ALT (SGPT) ≤ 2.5 X institutional upper limit of normal. Patients with confirmed liver metastases are permitted to have AST/ALT at levels ≤ 5X the institutional upper limit of normal.
  * Creatinine ≤ 1.5 X the institutional upper limit of normal.
  * Total cholesterol < 300 mg/dL
  * Triglycerides < 250 mg/dL
* The effects of everolimus on the developing human fetus are unknown. For this reason and because anti-neoplastic agents are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.
* Participants who achieve either a partial response or stable disease ≥ 4 months must agree to undergo a tumor biopsy, if safe and feasible, at the time of progressive disease while on study drug everolimus.

Exclusion Criteria:Participants who exhibit any of the following conditions at screening will not be eligible for admission into the study.

* Participants who have had any of the following:
* chemotherapy in the previous 2 weeks (6 weeks for nitrosoureas or mitomycin C)
* radiotherapy within 3 weeks
* investigational agents within 3 weeks prior to entering the study
* patients who have not recovered from significant (in the opinion of the investigator) adverse events due to previous agents administered.
* Child-Pugh B or C hepatic impairment. Patients with a history of hepatitis or significant exposure risk should be tested for hepatitis B and C with serologic markers: HBsAg, HBs Ab, HBcoreIgG Ab, HCV Ab. Patients with active hepatitis B or C are excluded.
* Any prior exposure to any PI3 kinase or mTOR inhibitor agent.
* Participants may not be receiving any other research study agents.
* Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases. Asymptomatic or treated brain metastases are acceptable.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to everolimus.
* A list of prohibited medications on study are listed in Section 5.5
* Chronic treatment with corticosteroids or other immunosuppressive therapy.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because everolimus has the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with everolimus, breastfeeding should be discontinued if the mother is treated with everolimus. These potential risks may also apply to other agents used in this study.
* Individuals with a recent history of a different malignancy are ineligible except for the following circumstances: 1) Individuals with a history of other malignancies are eligible if they have been disease-free for at least 3 years OR are deemed by the investigator to be at low risk for recurrence of that malignancy; 2) Individuals with the following cancers are eligible if diagnosed and treated within the past 3 years: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin.
* Individuals with known HIV infection are excluded from this study as combination antiretroviral therapy could potentially result in significant pharmacokinetic interactions with everolimus. In addition, these individuals are at increased risk of lethal infections due to the immunosuppressive effects of mTOR inhibition.
* Patients who have received live attenuated vaccines within 1 week of start of Everolimus. Patient should also avoid close contact with others who have received live attenuated vaccines. Examples of live attenuated vaccines include intranasal influenza, measles, mumps, rubella, oral polio, BCG, yellow fever, varicella and TY21a typhoid vaccines.
* Uncontrolled diabetes mellitus as defined by HbA1c >8% despite adequate therapy. Patients with a known history of impaired fasting glucose or diabetes mellitus (DM) may be included, however blood glucose and antidiabetic treatment must be monitored closely throughout the trial and adjusted as necessary.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-09; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Kwiatkowski, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Everolimus: Everolimus
  * Fixed doses orally once a day per each 28 day cycle
  * Participants will stay on study as long as they do not progress for a maximum of 24 months.
  * Tumor assessments will be performed after every 2 cycles for as long as they are on study.
  Everolimus
Period: Overall Study
Arm/Group | Everolimus
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Everolimus
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 14
Age, Continuous [Median (Full Range); unit: years] | 61.5 [43 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 25
  More than one race | 1
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 30
ECOG Performance Status [Median (Full Range); unit: units on a scale] — This is ECOG Performance Status 0 is the best, meaning in very good condition. 4 is the worse, meaning in very poor condition.
  units on a scale | 1 [0 to 1]

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: RECIST 1.1 criteria for Objective Response:
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by scan: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Baseline, Every 8 weeks, 2 Years
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus
Number analyzed (Participants) | 30
Participants | 2

2. Secondary Outcome: Duration of Response
Description: Duration of Response Rate
Time Frame: Baseline, Every 8 weeks, 2 Years
Population: Subjects with Partial Response
Measure: Median (Full Range); unit: months
Arm/Group | Everolimus
Number analyzed (Participants) | 2
months | 12.7 [4.8 to 20.7]

3. Secondary Outcome: Progression-free Survival
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Baseline, Up to 2 Years
Measure: Median (Full Range); unit: months
Arm/Group | Everolimus
Number analyzed (Participants) | 30
months | 2.0 [0.4 to 20.7]

4. Secondary Outcome: Overall Survival
Description: Overall Survival Rate
Time Frame: 4 Years
Measure: Median (Full Range); unit: months
Arm/Group | Everolimus
Number analyzed (Participants) | 30
months | 7.27 [0.43 to 39.93]

5. Secondary Outcome: Toxicity Rate
Description: CTCAE v4.0 Toxicity Rate Grade 3 or higher
Time Frame: 2 Years
Measure: Count of Participants; unit: Participants
Arm/Group | Everolimus
Number analyzed (Participants) | 30
Participants | 3

ADVERSE EVENTS:
Time Frame: 2 months after study discontinuation, up to 5 years
Description: National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE v4.0)
Arm/Group | Everolimus
All-Cause Mortality (participants affected / at risk) | 1/30
Serious Adverse Events (participants affected / at risk) | 3/30
Other Adverse Events (participants affected / at risk) | 20/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Everolimus (N=30)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Everolimus (N=30)
any adverse event per CTCAE v4.0 (Respiratory, thoracic and mediastinal disorders) | 20 (100) — any adverse event per CTCAE v4.0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-13): https://cdn.clinicaltrials.gov/large-docs/12/NCT02201212/Prot_SAP_000.pdf